CLINICAL TRIAL: NCT06703736
Title: Misure di funzionalità e deformità Dell'Apparato Muscolo-scheletrico Come "Biomarkers" Per il Trattamento di Malattie Ortopediche/Accessible Measurements of Mobility and Deformity as Biomarkers for Orthopaedic Treatments
Brief Title: Functional and Morphological Characterization of Multiple Osteochondromas Disorder
Acronym: MAMBO
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 333/2024/Sper/IOR
Record Dates: First submitted 2024-10-22; First posted 2024-11-25 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hereditary Multiple Osteochondromas
Keywords: Multiple osteochondromas; Functional limitation; Skeletal deformity; Gait analysis; IMU; Anthropometry; 3D scanning; Rare skeletal disease; Cartilage; Growth plates
MeSH Terms: conditions — Exostoses, Multiple Hereditary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple osteochondromas patients: The cohort is composed of patients suffering from hereditary multiple osteochondromas (HMO) and it contains 30 subjects: 15 minors (6-17 years) and 15 adults (18-40 years). The inclusion criteria of HMO cohort are: clinical and/or molecular diagnosis of Multiple Osteochondromas; male and female subjects; collection of appropriate informed consent; ability to walk a linear path without aids; presence of OM localized at lower limbs; ability to undergo all procedures required by the protocol. Are excluded from the cohort subjects with body mass index (BMI) equal to or greater than 30.
- Healthy subjects: Healthy subjects are control population, equivalent in gender and age to the investigated population. The cohort is composed of 30 subjects: 15 minors (6-17 years) and 15 adults (18-40 years).The inclusion criteria of healthy cohort are: absence of neuro-muskuloskeletal or other limb-limiting conditions in the lower limbs; male and female subjects; collection of appropriate informed consent; ability to undergo all procedures required by the protocol. Are excluded from the cohort subjects with body mass index (BMI) equal to or greater than 30.

SUMMARY:
The main purpose of the study is the characterization of functional and morphological alterations due to multiple osteochondromas in a pediatric and adult population through the identification of relevant anthropometric and functional parameters. The morphological and functional data, supplemented with clinical and postural data, will allow the characterization of the disease with an holistic approach that can provide important information to properly assess timing for surgical treatments and to improve the quality of life of these patients. Another goal of the study is the assessment and the validation of novel instruments and tools to measure joint mobility and bone deformity. These instruments should be easy-to-use and designed to be operated locally by the patients themselves and/or in small clinics by operators with little training and no specific high-technical knowledge. The final goal of the study is the assessment of the quality of life and balance perception of patients, using questionnaires.

DETAILED DESCRIPTION:
Hereditary Multiple Osteochondromas (HMO) disease, also known as 'Hereditary Multiple Exostosis', is a rare autosomal dominant musculoskeletal disorder whose prevalence is estimated at 1:50000. It is characterised by benign osteo-cartilaginous tumours called 'osteochondromas' or 'exostoses', cartilage capped bony outgrowths that originate from the perichondrium of long bones and from the surface of flat bones. The development and growth of exostoses occur in parallel with the growth of the subject and then stop at skeletal maturity. HMO is characterized by phenotypic heterogeneity and the most important complication is malignant transformation of osteochondroma towards secondary peripheral chondrosarcoma, which is estimated to occur in 0.5-5%. In most case, the disease is characterized by a broad-spectrum of mutations in the EXT1 and EXT2 genes coding for transmembrane glycoproteins with glycosyl-transferase activity.

Patients with HMO are subject to functional and postural alterations of the musculoskeletal system caused by bone deformities that begin to appear at an early age. The characterization and monitoring of residual mobility is essential to objectively quantify the motor and morphological deficit and to understand the mechanisms of action and evolution of this pathology. To date, there are no studies in the literature on the instrumental characterisation of OM. Furthermore, although skeletal structure deformities are one of the main causes of functional alterations, studies on the description and instrumental characterisation of macroscopic morphological alterations are limited. The expected results are morphological data (shape, position, size and numerosity) of osteochondromas and functional data (range of motion of the joints affected by the pathology). Other expected results are: accuracy and repeatability of the instruments to be used for monitoring pathology; an overall evaluation of the experience by means of an evaluation questionnaire; information on the feasibility of the pilot study for the implementation of a study on a larger cohort; identification of new prevention and treatment strategies in patients with rare diseases clinically similar to OM (e.g. metachondromatosis) or for other skeletal diseases that are not rare but widespread (e.g. osteoarthritis).

ELIGIBILITY:
Inclusion Criteria:

For multiple osteochondromas cohort inclusion criteria are:

* clinical and/or molecular diagnosis of Multiple Osteochondromas;
* male and female subjects;
* age minors: 6-17 years at enrollment and adult age: 18-40 years at enrollment;
* collection of appropriate informed consent;
* ability to walk a linear path without aids;
* presence of multiple osteochondromas localized at lower limbs;
* ability to undergo all procedures required by the protocol.

For healthy cohort inclusion criteria are:

* absence of neuro-muskuloskeletal or other limb-limiting conditions in the lower limbs;
* male and female subjects;
* age minors: 6-17 years at enrollment and adult age: 18-40 years at enrollment;
* collection of appropriate informed consent;
* ability to undergo all procedures required by the protocol.

Exclusion Criteria:

* Persons who do not fit the inclusion criteria;
* Any reason which, in the opinion of the investigator, would result in the inability of the participant to comply with the protocol.
* BMI equal to or greater than 30.

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The multiple osteochondromas population is selected from patients taken over by CeMaRS (Centre of Rare Skeletal Disorders) of Istituto Ortopedico Rizzoli (IOR), while the healthy population is recruit via social and IOR website, possibly including healthy relatives of recruited patients if the absence of the causative genetic variant of the disease and the absence of its clinical manifestations are proven.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Functional motor assessment | From subjects enrollment to the end of the assessment. Patients repeat these activities after 12 months from the first evaluation, while healthy subjects carry out the same activities of unhealthy population only once.
  Analysis of the following motor tasks is executed: planar linear walking, overcoming a step/obstacle, standing up/ sitting down from a chair. Analysis of these movements includes:
  1. joint kinematics obtained through inertial sensors (IMU) that are attached to the body segments by means of bands or double-sided tape;
  2. joint kinetics (joint torque and powers) obtained from ground reaction force data, measured with the force platforms on the laboratory floor and from joint kinematics;
  3. plantar pressure maps by means of a baropodometric platform positioned on the laboratory floor that will measure plantar pressure data in static and dynamic.
Anthropometric parameters assessment | From subjects enrollment to the end of the assessment. Patients repeat these activities after 12 months from the first evaluation, while healthy subjects carry out the same activities of unhealthy population only once.
  Body measurement using 3D scanning is carried out. The subject should wear underwear or short and tight clothing. The subject should remain as still as possible in a standing position while being scanned.

SECONDARY OUTCOMES:
Evaluation of experimental protocols using simplified instrumentation | through study completion
  The analysis of kinematic parameters will be carried out with a gold standard stereophotogrammetric instrument and by means of wearable IMU sensor. The analysis of anthropometric parameters will be carried out by means of a high resolution manual 3D scanning system (slower but more accurate), and by means of a low resolution 3D scanning system without operator intervention (faster but less accurate). The comparison between the two instruments will allow optimisation of the acquisition parameters and establish the reliability and accuracy of ad-hoc assessment protocols for monitoring patients.
Evaluation questionnaire | The questionnaire is administered to the cohort of patients at the first acquisition and at 12-month follow-up.
  The questionnaire aims to collect opinions on the experience lived during the execution of the motor tasks and other planned activities so as to be able to assess the opinion of the multiple osteochondromas participants in terms of feasibility and also to identify areas for improvement to carry out a study with a wider range of case studies.
Assessment of quality of life and balance perception of hereditary multiple osteochondromas patients | through study completion
  This secondary outcome assessment involves only the cohort of hereditary multiple osteochondromas subjects and not the healthy ones. Questionnaires concerning quality of life (EuroQol-5) and perceived sense of balance (ABC scale) will be administered to each subject.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided